CLINICAL TRIAL: NCT03004703
Title: ASSessing the Effect of Anti-IL-6 Treatment in Myocardial Infarction: The ASSAIL-MI Trial
Acronym: ASSAIL-MI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lars Gullestad, Profesor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASSAIL-MI 2.0; 2016-002581-31 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: Interleukin 6; Tocilizumab; Acute coronary syndrome; STEMI; Inflammation
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Inflammation | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug (Experimental): Tocilizumab, 20 mg/ml; 14 ml (280 mg) dissolved in 100 ml NaCl 0.9 % i.v. once.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): Sodium chloride 0.9%; 100 ml i.v. once.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Tocilizumab — Active drug: Tocilizumab, 20 mg/ml; 14 ml (280 mg) dissolved in 100 ml NaCl 0.9 % i.v. once.
  Other Names: RoActemra®,
  Arms: Active drug
Drug: Sodium chloride 0.9% — Placebo: Sodium chloride 0.9%; 100 ml i.v. once.
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
The main goal of this study is to evaluate the ability of a single administration of tocilizumab to reduce myocardial damage in patients presenting with an acute ST-segment elevation myocardial infarction (STEMI). Secondary objectives are to assess the impact of treatment on: (i) final infarct size, (ii) left ventricular size and function, (iii) inflammation, (iv) extracellular matrix remodeling, (v) lipid parameters, (vi) platelet activation and additional pro- and anti-thrombotic parameters, and (vii) study drug safety and tolerability.

DETAILED DESCRIPTION:
Myocardial infarction (MI) is a major contributor to morbidity and mortality in the Western world. The main determinant of death and complications is infarct size, and limitation of the infarct size has therefore been an important objective for strategies to improve outcome. In patients presenting with an acute ST segment elevation myocardial infarction (STEMI), urgent myocardial reperfusion with percutaneous coronary intervention (PCI) is the most effective treatment to this end. However, despite PCI, the morbidity and mortality in patients with STEMI remain substantial. This fact suggests that other, adjuvant strategies are required to reduce infarct size and improve outcome. The inflammatory cytokine interleukin (IL)-6 is an important mediator of plaque destabilisation and rupture in acute coronary syndrome (ACS) and may contribute to the ischemia-reperfusion injury succeeding revascularisation. Experimental studies suggest that IL-6 inhibition can limit infarct size through anti-inflammatory mechanisms.(ref)

The investigators recently conducted a double blind, placebo controlled trial in 117 patients with non-ST segment elevation myocardial infarction (NSTEMI) who presented within 72 hour after the onset of chest pain. In this study, a single, intravenous dose of the IL-6 antagonist tocilizumab reduced the inflammatory activity by more than 50% in the days subsequent to the intervention. Importantly, tocilizumab also reduced troponin T (TnT) levels, suggesting that patients receiving tocilizumab sustained less myocardial damage than patients who received placebo.1

Interleukin-6 inhibition might limit infarct size through reduced myocardial inflammation, but theoretically, it could also inhibit the repair process within the injured area. While the recent study suggests that IL-6 inhibition has largely favourable effects in NSTEMI, it remains to be seen if similar, beneficial effects can be obtained in patients with STEMI. On this background, the investigators want to investigate the effect of tocilizumab in patients with acute STEMI. The postulate is that a single dose of tocilizumab (RoActemra®) will have favourable effects on infarct size, as assessed by markers of myocardial necrosis and cardiac magnetic resonance imaging (CMR), without negative consequences for the repair process in these patients. The hypothesis will be tested in a randomised, double blind, placebo controlled trial comprising 200 patients with acute STEMI.

This is a phase 2 study on a new and exciting anti-inflammatory strategy in cardiovascular disease. It will be conducted at three experienced, high volume centres in Norway, and will target new and yet unmodified mechanisms during myocardial infarction. The ambition is to improve the prognosis of patients with ACS, with potential to change clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients will be screened for eligibility upon admittance due to acute STEMI at either participating site. All of the following conditions must apply to the prospective patient at screening prior to receiving study agent:

* New ST elevation at the J-point in two contiguous leads (cut-points: 0.2mV in men and >0.15 mV in women in leads V2-V3 and/or >0.1 mV in other leads) in combination with symptoms consistent with acute MI.
* Presentation within 6 hours of chest pain.
* Indication for urgent coronary angiography with intent to reperfuse presumed occluded vessel.
* Age between 18 and 80 years.
* Informed consent obtained and documented according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* NSTEMI (non-ST segment elevation in ECG).
* Left bundle branch block in ECG
* History of previous MI
* Cardiogenic shock.
* Fibrinolytic therapy within 72 hours prior to admission.
* Cardiac arrest / ventricular fibrillation.
* History of severe renal failure with estimated glomerular filtration rate < 30 ml/minutes.
* Known, current liver disease
* History of concurrent inflammatory, biliary obstructive or malignant disease
* A history of chronic or concurrent infectious disease, including a history of HIV, tuberculosis, or hepatitis B or C.
* Known, uncontrolled lower gastrointestinal (GI) disease such as diverticulitis, Crohn's disease, ulcerative colitis, or other symptomatic lower GI conditions that could predispose to GI perforations
* Major surgery within 8 weeks prior or after baseline
* History of central nervous system demyelinating or seizure disorders
* History of primary or secondary immunodeficiency
* Treatment with immunosuppressants other than low dose corticosteroids (equivalent to 5 mg of prednisone or less) at the time of randomisation
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or to tocilizumab
* Other contraindications to study medication
* Pregnancy, possible pregnancy or breast-feeding - women of child-bearing potential or breastfeeding mothers cannot participate. A woman is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Contraindications to CMR (pacemaker, CRT, ICD, certain ferromagnetic implants, severe claustrophobia, allergy to contrast medium).
* Any condition/circumstances believed to interfere with the ability to comply with protocol.
* Any reason why, in the opinion of the investigator, the patient should not participate.
* Failure to obtain written, informed consent by patient or next of kin, for instance in case of patient death after consent has been provided in oral.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the between-group difference in the myocardial salvage index as measured in the acute phase by cardiac magnetic resonance (CMR) imaging with late gadolinium enhancement (LGE). | 6 months

SECONDARY OUTCOMES:
The between-group difference in the AUC for Troponin T (TnT) during index hospitalisation | 24 -72 hours after randomisation
The extent of microvascular obstruction as measured by CMR after 3 - 7 days | 3 - 7 days after randomisation
Final infarct size as measured by CMR 6 months after randomisation | 6 months after randomisation
Left ventricular size as assessed by CMR 6 months after randomisation | 6 months after randomisation
Baseline-adjusted NT-proBNP at 6 months after randomisation | 6 months after randomisation
The AUC of Creatine Kinase-MB (CK-MB) during index hospitalisation | 24-72 hours after randomisation
The AUC of C-reactive protein (CRP) during index hospitalisation | 24-72 hours after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, Professor, MD, PhD, Principal Investigator — Oslo University Hospital; Bjørn Bendz, Associate Professor, MD, PhD, Study Chair — Oslo University Hospital; Pål Aukrust, Professor, MD, PhD, Study Chair — Oslo University Hospital; Svend Aakhus, Professor, MD, PhD, Study Chair — Oslo University Hospital; Rune Wiseth, Professor, MD, PhD, Study Chair — St. Olavs Hospital; Jan Kristian Damaas, Professor, MD, PhD, Study Chair — St. Olavs Hospital; Geir Øystein Andersen, MD, PhD, Study Chair — Oslo University Hospital, Ullevål; Nils Einar Kløw, Professor, MD, PhD, Study Chair — Oslo University Hospital, Ullevål; Anders Opdahl, MD, PhD, Study Chair — Oslo University Hospital, Ullevål
Locations (3):
- Norway (3):
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevål, Oslo
  - St. Olav Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Kleveland O, Kunszt G, Bratlie M, Ueland T, Broch K, Holte E, Michelsen AE, Bendz B, Amundsen BH, Espevik T, Aakhus S, Damas JK, Aukrust P, Wiseth R, Gullestad L. Effect of a single dose of the interleukin-6 receptor antagonist tocilizumab on inflammation and troponin T release in patients with non-ST-elevation myocardial infarction: a double-blind, randomized, placebo-controlled phase 2 trial. Eur Heart J. 2016 Aug 7;37(30):2406-13. doi: 10.1093/eurheartj/ehw171. Epub 2016 May 8. PMID 27161611
- [Background] Braunwald E, Kloner RA. Myocardial reperfusion: a double-edged sword? J Clin Invest. 1985 Nov;76(5):1713-9. doi: 10.1172/JCI112160. No abstract available. PMID 4056048
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Background] Libby P. Molecular bases of the acute coronary syndromes. Circulation. 1995 Jun 1;91(11):2844-50. doi: 10.1161/01.cir.91.11.2844. No abstract available. PMID 7758192
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Hou T, Tieu BC, Ray S, Recinos Iii A, Cui R, Tilton RG, Brasier AR. Roles of IL-6-gp130 Signaling in Vascular Inflammation. Curr Cardiol Rev. 2008 Aug;4(3):179-92. doi: 10.2174/157340308785160570. PMID 19936194
- [Background] Ritschel VN, Seljeflot I, Arnesen H, Halvorsen S, Eritsland J, Fagerland MW, Andersen GO. Circulating Levels of IL-6 Receptor and gp130 and Long-Term Clinical Outcomes in ST-Elevation Myocardial Infarction. J Am Heart Assoc. 2016 Jun 13;5(6):e003014. doi: 10.1161/JAHA.115.003014. PMID 27412895
- [Background] Piot C, Croisille P, Staat P, Thibault H, Rioufol G, Mewton N, Elbelghiti R, Cung TT, Bonnefoy E, Angoulvant D, Macia C, Raczka F, Sportouch C, Gahide G, Finet G, Andre-Fouet X, Revel D, Kirkorian G, Monassier JP, Derumeaux G, Ovize M. Effect of cyclosporine on reperfusion injury in acute myocardial infarction. N Engl J Med. 2008 Jul 31;359(5):473-81. doi: 10.1056/NEJMoa071142. PMID 18669426
- [Background] Granger CB, Mahaffey KW, Weaver WD, Theroux P, Hochman JS, Filloon TG, Rollins S, Todaro TG, Nicolau JC, Ruzyllo W, Armstrong PW; COMMA Investigators. Pexelizumab, an anti-C5 complement antibody, as adjunctive therapy to primary percutaneous coronary intervention in acute myocardial infarction: the COMplement inhibition in Myocardial infarction treated with Angioplasty (COMMA) trial. Circulation. 2003 Sep 9;108(10):1184-90. doi: 10.1161/01.CIR.0000087447.12918.85. Epub 2003 Aug 18. PMID 12925454
- [Background] Deftereos S, Giannopoulos G, Angelidis C, Alexopoulos N, Filippatos G, Papoutsidakis N, Sianos G, Goudevenos J, Alexopoulos D, Pyrgakis V, Cleman MW, Manolis AS, Tousoulis D, Lekakis J. Anti-Inflammatory Treatment With Colchicine in Acute Myocardial Infarction: A Pilot Study. Circulation. 2015 Oct 13;132(15):1395-403. doi: 10.1161/CIRCULATIONAHA.115.017611. Epub 2015 Aug 11. PMID 26265659
- [Background] Biasillo G, Leo M, Della Bona R, Biasucci LM. Inflammatory biomarkers and coronary heart disease: from bench to bedside and back. Intern Emerg Med. 2010 Jun;5(3):225-33. doi: 10.1007/s11739-010-0361-1. Epub 2010 Feb 25. PMID 20182820
- [Background] Kinlay S, Schwartz GG, Olsson AG, Rifai N, Leslie SJ, Sasiela WJ, Szarek M, Libby P, Ganz P; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering Study Investigators. High-dose atorvastatin enhances the decline in inflammatory markers in patients with acute coronary syndromes in the MIRACL study. Circulation. 2003 Sep 30;108(13):1560-6. doi: 10.1161/01.CIR.0000091404.09558.AF. Epub 2003 Sep 15. PMID 12975259
- [Background] Oldfield V, Dhillon S, Plosker GL. Tocilizumab: a review of its use in the management of rheumatoid arthritis. Drugs. 2009;69(5):609-32. doi: 10.2165/00003495-200969050-00007. PMID 19368420
- [Background] Eitel I, de Waha S, Wohrle J, Fuernau G, Lurz P, Pauschinger M, Desch S, Schuler G, Thiele H. Comprehensive prognosis assessment by CMR imaging after ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2014 Sep 23;64(12):1217-26. doi: 10.1016/j.jacc.2014.06.1194. PMID 25236513
- [Background] Erlinge D, Gotberg M, Lang I, Holzer M, Noc M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Harnek J, Olivecrona GK. Rapid endovascular catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. The CHILL-MI trial: a randomized controlled study of the use of central venous catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. J Am Coll Cardiol. 2014 May 13;63(18):1857-65. doi: 10.1016/j.jacc.2013.12.027. Epub 2014 Feb 5. PMID 24509284
- [Background] Atar D, Arheden H, Berdeaux A, Bonnet JL, Carlsson M, Clemmensen P, Cuvier V, Danchin N, Dubois-Rande JL, Engblom H, Erlinge D, Firat H, Halvorsen S, Hansen HS, Hauke W, Heiberg E, Koul S, Larsen AI, Le Corvoisier P, Nordrehaug JE, Paganelli F, Pruss RM, Rousseau H, Schaller S, Sonou G, Tuseth V, Veys J, Vicaut E, Jensen SE. Effect of intravenous TRO40303 as an adjunct to primary percutaneous coronary intervention for acute ST-elevation myocardial infarction: MITOCARE study results. Eur Heart J. 2015 Jan 7;36(2):112-9. doi: 10.1093/eurheartj/ehu331. Epub 2014 Sep 1. PMID 25179768
- [Background] Ibanez B, Macaya C, Sanchez-Brunete V, Pizarro G, Fernandez-Friera L, Mateos A, Fernandez-Ortiz A, Garcia-Ruiz JM, Garcia-Alvarez A, Iniguez A, Jimenez-Borreguero J, Lopez-Romero P, Fernandez-Jimenez R, Goicolea J, Ruiz-Mateos B, Bastante T, Arias M, Iglesias-Vazquez JA, Rodriguez MD, Escalera N, Acebal C, Cabrera JA, Valenciano J, Perez de Prado A, Fernandez-Campos MJ, Casado I, Garcia-Rubira JC, Garcia-Prieto J, Sanz-Rosa D, Cuellas C, Hernandez-Antolin R, Albarran A, Fernandez-Vazquez F, de la Torre-Hernandez JM, Pocock S, Sanz G, Fuster V. Effect of early metoprolol on infarct size in ST-segment-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention: the Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction (METOCARD-CNIC) trial. Circulation. 2013 Oct 1;128(14):1495-503. doi: 10.1161/CIRCULATIONAHA.113.003653. Epub 2013 Sep 3. PMID 24002794
- [Background] Eitel I, Stiermaier T, Rommel KP, Fuernau G, Sandri M, Mangner N, Linke A, Erbs S, Lurz P, Boudriot E, Mende M, Desch S, Schuler G, Thiele H. Cardioprotection by combined intrahospital remote ischaemic perconditioning and postconditioning in ST-elevation myocardial infarction: the randomized LIPSIA CONDITIONING trial. Eur Heart J. 2015 Nov 21;36(44):3049-57. doi: 10.1093/eurheartj/ehv463. Epub 2015 Sep 17. PMID 26385956
- [Background] Galderisi M, Henein MY, D'hooge J, Sicari R, Badano LP, Zamorano JL, Roelandt JR; European Association of Echocardiography. Recommendations of the European Association of Echocardiography: how to use echo-Doppler in clinical trials: different modalities for different purposes. Eur J Echocardiogr. 2011 May;12(5):339-53. doi: 10.1093/ejechocard/jer051. PMID 21555455
- [Background] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Gibbons RJ, Valeti US, Araoz PA, Jaffe AS. The quantification of infarct size. J Am Coll Cardiol. 2004 Oct 19;44(8):1533-42. doi: 10.1016/j.jacc.2004.06.071. PMID 15489082
- [Background] Engblom H, Heiberg E, Erlinge D, Jensen SE, Nordrehaug JE, Dubois-Rande JL, Halvorsen S, Hoffmann P, Koul S, Carlsson M, Atar D, Arheden H. Sample Size in Clinical Cardioprotection Trials Using Myocardial Salvage Index, Infarct Size, or Biochemical Markers as Endpoint. J Am Heart Assoc. 2016 Mar 9;5(3):e002708. doi: 10.1161/JAHA.115.002708. PMID 26961520
- [Derived] Kindberg KM, Broch K, Andersen GO, Anstensrud AK, Akra S, Woxholt S, Tollefsen IM, Ueland T, Amundsen BH, Klow NE, Halvorsen B, Dahl TB, Huse C, Murphy SL, Damas JK, Opdahl A, Wiseth R, Gullestad L, Aukrust P, Santos-Gallego C, Seljeflot I, Stokke MK, Helseth R. Neutrophil Extracellular Traps in ST-Segment Elevation Myocardial Infarction: Reduced by Tocilizumab and Associated With Infarct Size. JACC Adv. 2024 Aug 15;3(9):101193. doi: 10.1016/j.jacadv.2024.101193. eCollection 2024 Sep. PMID 39247678
- [Derived] Woxholt S, Ueland T, Aukrust P, Anstensrud AK, Broch K, Tollefsen IM, Ryan L, Bendz B, Hopp E, Klow NE, Seljeflot I, Halvorsen B, Dahl TB, Huse C, Andersen GO, Gullestad L, Wiseth R, Amundsen BH, Damas JK, Kleveland O. Cytokine pattern in patients with ST-elevation myocardial infarction treated with the interleukin-6 receptor antagonist tocilizumab. Open Heart. 2023 Aug;10(2):e002301. doi: 10.1136/openhrt-2023-002301. PMID 37591633
- [Derived] Broch K, Anstensrud AK, Woxholt S, Sharma K, Tollefsen IM, Bendz B, Aakhus S, Ueland T, Amundsen BH, Damas JK, Berg ES, Bjorkelund E, Bendz C, Hopp E, Kleveland O, Stensaeth KH, Opdahl A, Klow NE, Seljeflot I, Andersen GO, Wiseth R, Aukrust P, Gullestad L. Randomized Trial of Interleukin-6 Receptor Inhibition in Patients With Acute ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2021 Apr 20;77(15):1845-1855. doi: 10.1016/j.jacc.2021.02.049. PMID 33858620
- [Derived] Anstensrud AK, Woxholt S, Sharma K, Broch K, Bendz B, Aakhus S, Ueland T, Amundsen BH, Damas JK, Hopp E, Kleveland O, Stensaeth KH, Opdahl A, Klow NE, Seljeflot I, Andersen GO, Wiseth R, Aukrust P, Gullestad L. Rationale for the ASSAIL-MI-trial: a randomised controlled trial designed to assess the effect of tocilizumab on myocardial salvage in patients with acute ST-elevation myocardial infarction (STEMI). Open Heart. 2019 Oct 15;6(2):e001108. doi: 10.1136/openhrt-2019-001108. eCollection 2019. PMID 31673391